CLINICAL TRIAL: NCT04748484
Title: Clinical Evaluation of the Medical Device (MD) (Caloprothese Connected Kit, CCK)- Comprising a Sleeve and a Sock - in Amputees Suffering From Rebellious Neuropathic Pain on the Residual Limb and / or Phantom Limb
Brief Title: Clinical Evaluation of the Medical Device (MD) (Caloprothese Connected Kit, CCK)
Acronym: KCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gregand Innovations (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-A00396-33
Record Dates: First submitted 2021-01-11; First posted 2021-02-10 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Neuropathic Pain; Phantom Limb Pain
Keywords: phantom limb pain; SCED; medical device
MeSH Terms: conditions — Neuralgia; Phantom Limb

STUDY DESIGN:
Intervention Model Description: Single case experimental design : the principle is to evaluate intensively and prospectively a small group of subjects, each case being its own comparator
Masking Description: The medical device will be active or inactive, but the patient nor the investigator won't know if the medical device is active or not. The battery charge indicator will work the same whether the device is operating or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- KCC active or inactive (Other): The medical device KCC will be active, or inactive. Randomization will define when and how long time the medical device will be active, and when and how long time the medical device will be inactive. The patient won't know if the medical device is active or not. The battery charge indicator will work the same whether the device is operating or not.
  Interventions: Device: KCC Active or inactive

INTERVENTIONS:
Device: KCC Active or inactive — Depending of the randomization, the KCC will be active or inactive, and will provide heat when active, but the patient won't know if the medical device is active or not. The battery charge indicator will work the same whether the device is operating or not.

SUMMARY:
Neuropathic pain is common in limb amputees and causes reductions in activity and participation as well as impaired quality of life. Some of these pains lead to the diagnosis of a responsible lesion and to precise and effective treatments (amputation neuroma pains, for example), whether they are etiological or symptomatic. Other pains of a neuropathic character remain totally or partially resistant to symptomatic treatment. Their appearance, intensity, duration and frequency vary depending on the amputee.

Old scientific data confirmed by modern imagery indicates a process of reorganization of cortical areas by multimodal afferents. This reconstruction, coherent or not of the body diagram, is at the genesis of sensations, normal or not, in the amputee.

Early plurimodal reassignment constitutes the founding principle of the rehabilitation of amputees: tactile afferents, visual afferents, motor afferents, proprioceptive afferents. Rehabilitation techniques and early fitting contribute to this reafferentation and to the functional integration of the fitting and to the quality of life of the amputee.

Scientific work by Katz et al, and experiences of amputees relieved by the application of local heat or stay in hot climatic zones show that the thermoregulation of the residual limb could be of interest.

It has been shown that these pain conditions are often related to a reduction in superficial blood flow to the distal part of the stump. The physiological response of the body to variations in outside temperature physiologically consists in the regulation of skin temperature. The goal seems to keep the body in a so-called "thermal neutrality" zone, substantially between 30 ° C and 33 ° C, by vasodilation or vasoconstriction of the superficial blood vessels depending on exposure to cold or heat.

An innovative medical device has been developed for a regulated thermal re-afferentation of the residual limb, during and outside the wearing of the prosthesis. The Connected Caloprosthesis Kit (CCK®) includes a connected sleeve put in place when wearing the prosthesis (interface between the skin and the socket) and a connected sock to put in place outside of wearing the prosthesis. These 2 devices include an autonomous heating and regulation process, which maintains the amputation stump in the area known as "skin thermal normality". This device is non-invasive. It includes a silicone sleeve and a heating sock for femoral or tibial amputee patients equipped with an expandable textile warmer, a flexible micro-temperature sensor and a 4-conductor extensible cable connected to a thermoregulation box worn as a belt which regulates the temperature of the stumps in the thermal neutrality zone between 30 and 33°C.

In order to assess the therapeutic effect of CCK®, given the heterogeneity of the population and the small number of patients eligible for the study, the Single Case Experimental Design (multiple baselines design) seems to us to be the methodology the most suitable: the principle is to evaluate intensively and prospectively a small group of subjects, each case being its own comparator. The methodology is defined a priori including systematic observations and repeated measurements at a defined frequency before, during, or even after the intervention introduced in a sequential and randomized manner. The data analysis can be individual and therefore patient-specific, but also group with the calculation of the size of the therapeutic effect and the calculation of significance.

This design therefore makes it possible to overcome the difficulties encountered during randomized controlled trials: having to have a large number of subjects necessary to show a significant difference in the medical device and to have a homogeneous population.

This methodology is therefore not a description of a clinical case but an alternative methodology to randomized controlled trials. In fact, it is considered by the Oxford Center for Evidence-Based Medicine 2011 to be level I, like the randomized controlled trials.

The proposed clinical study therefore has a dual objective: practical as a new treatment therapy by validating this medical device and theoretical, supporting the pathogenic model of painful sensations in amputees

ELIGIBILITY:
Inclusion Criteria:

* Patient seen in consultation motivated by residual limb pain
* Adult with background pain (Lickert scale ≥ 5/10) or with pain attacks (Lickert scale ≥ 5/10) whose frequency is more than once per week
* Patient with a DN4 score > 4/10 (Score validated in neuropathic pain)
* Patient with trans-femoral or trans-tibial amputation
* Patient whose amputation was over 1 year ago regardless of the aetiology of his amputation.

Exclusion Criteria:

Patient :

* under 18 year old
* With a silicone allergy
* Usually fitted by means of suspension by a seal in sleeve, by suspension by vacuum pump requiring a polyurethane sleeve
* Presenting any pathology of the stump explaining the pain on clinical arguments, complemented if necessary by additional investigations: neuroma, bone or vascular pathology or conflicts with the socket…
* With bilateral lower limb amputation
* Not being able to use a Smartphone
* Not wishing to participate in the study
* Adult subject to legal protection or unable to express consent
* Pregnant or breastfeeding females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Intensity of the overall pain (background pain and paroxysmal pain) on 0-10 numerical scale | Up to 5 months
  The primary judgment criteria will be the evaluation of the intensity of the overall pain (background pain and paroxysmal pain) on 0-10 numerical scale over the last 48 hours measured three times a week during the follow up of the patient

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Hôpital d'Instruction des Armées Percy -, Clamart
  - Irr Nancy, Nancy
  - CRF La Tourmaline, Saint-Herblain
  - Institut Universitaire de Réadaptation Clemenceau, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided